CLINICAL TRIAL: NCT02736552
Title: A Prospective,Multicentral,Open-label,Randomized,Controlled,Phase III Clinical Trial to Compare S-1 for 6 Months to 1 Year as Adjuvant Chemotherapy After D2 Resection in Patients With Gastric Cancer Staged II , IIIA or IIIB.
Brief Title: Compare S-1 for 6 Months to 1 Year as Adjuvant Chemotherapy After D2 Resection in Patients With Gastric Cancer Staged II , IIIA or IIIB.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Anhui Provincial Hospital (Other Government); The First Affiliated Hospital of Anhui Medical University (Other); Anqing Municipal Hospital (Other); Yuebei People's Hospital (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shenzhen People's Hospital (Other); First Affiliated Hospital of Wannan Medical College (Other); Lishui hospital of Zhejiang University (Unknown); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGCG001
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Adjuvant chemotherapy; S-1; D2 resection
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-1 for 6 months (Experimental): S-1 80-120mg daily for 14 days in 3 weeks for totally 6 months after D2 resection
  Interventions: Drug: S-1 for 6 months
- S-1 for 1 year (Active Comparator): S-1 80-120mg daily for 14 days in 3 weeks for totally 1 year after D2 resection
  Interventions: Drug: S-1 for 1 year

INTERVENTIONS:
Drug: S-1 for 6 months — 6 months S-1 after D2 resection
  Arms: S-1 for 6 months
Drug: S-1 for 1 year — 1 year S-1 after D2 resection
  Arms: S-1 for 1 year

SUMMARY:
The study aims to compare the efficacy and safety of S-1 for 6 months versus S-1 for 1 year as adjuvant chemotherapy after D2 resection in patients with gastric cancer.

Hypothesis: For gastric patients after D2 resection, S-1 for 6 months shows non-inferiority to S-1 for 1 year in disease free survival(DFS), overall survival (OS) and safety.

DETAILED DESCRIPTION:
It has been identified that S-1 is an effective adjuvant treatment for East Asian patients who have undergone a D2 dissection for locally advanced gastric cancer（GC) in the Japanese Adjuvant Chemotherapy Trial of TS-1（S-1) for Gastric Cancer (ACTS-GC) trail , And S-1 has become one of the standard therapies to these patients. But it is still unknown whether it would improve equally or even more to overall survival(OS) and disease free survival(DFS) than S-1 for 1 year compared with S-1 for 6 months. As a result , An further clinical trail is still needed, This trial is designed to investigate the efficacy and safety of S-1 for 6 months versus S-1 for 1 year as adjuvant chemotherapy after D2 resection in patients with gastric cancer.

In this study, patients histologically confirmed stage II, IIIA or IIIB and who received D2 resection were randomly assigned to receive S-1 for 6 months or S-1 for 1 year. Patients aged from 18 to 75 years and adequate organ function, are randomized 1:1 to S-1 for 6 months and S-1 for 1 year. Both are the 3-week recycle of S-1 (80-120mg per day) for 2 weeks ,followed by 1 week of rest. The primary end point is 3-year DFS, and secondary end point is 5-year OS and safety. Final study analysis will be conducted in the end of the 5th year after the last patient's enrollment.In summary, we hold the hypothesis that S-1 for 6 months is equally effective, safer, and easier to carry out. If possible, there will be a new adjuvant chemotherapy strategy for gastric cancer patients after D2 resection.

To ensure the quality of the study, two interim analyses will be planned at the half and the completion of the study respectively. The DATA and Safety Monitoring Committee will independently review the interim analysis and stop the study ahead of schedule if necessary. Furthermore, to improve the study progress and quality, the in-house interim monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 75 years old.
2. Be proven to be primary adenocarcinoma of gastric cancer and staged II，IIIA or IIIB by pathological evidences
3. R0 surgery with lymphadenectomy
4. Without any other malignancies
5. ECOG (ECOG score standard) performance status of 0 or 1 and expected to survive more than 6 months
6. No contraindications to chemotherapy, including normal peripheral blood routine, liver and kidney function and electrocardiogram （WBC≥4.0 x 109 /L, NEU≥1.5 x 109 /L,PLT≥100 x 109 /L and HGB≥90g/L).

Exclusion Criteria:

1. Female in pregnancy or lactation, or refuse to receive Contraception measures during chemotherapy.
2. Patients with stage I, IIIC and IV.
3. Unavailable for R0 resection and D2 lymph node dissection.
4. Suffering from other uncontrolled diseases, such as other tumors, acute and Chronic infection.
5. With severe heart disease, including: congestive heart failure, uncontrolled arrhythmias, unstable angina, myocardial infarction, severe heart valve disease and resistant hypertension.
6. Any Known or suspected history of drug allergy test.
7. The researchers believe the patient is not able to complete the entire course of the experiment.
8. Patients (within 4 weeks) are receiving any other anti-cancer drugs therapy, biological therapy, radiation therapy, or Immunosuppressive therapy.
9. Patients conform to any of the following: post-organ transplant, necessary for long-term immunosuppressive or suffering with autoimmune diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-year

SECONDARY OUTCOMES:
Overall survival | 5-year
Overall survival | 3-year
Side effects | 12 months
  Complications such as Nausea, vomiting, myelosuppression and Liver or kidney function disorder.

OTHER OUTCOMES:
Treatment expense | 12 months
  Total costs of treatment

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Cancer Center of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Lishui hospital of Zhejiang University, Lishui, Zhejiang

REFERENCES:
- [Background] Sasako M, Sakuramoto S, Katai H, Kinoshita T, Furukawa H, Yamaguchi T, Nashimoto A, Fujii M, Nakajima T, Ohashi Y. Five-year outcomes of a randomized phase III trial comparing adjuvant chemotherapy with S-1 versus surgery alone in stage II or III gastric cancer. J Clin Oncol. 2011 Nov 20;29(33):4387-93. doi: 10.1200/JCO.2011.36.5908. Epub 2011 Oct 17. PMID 22010012
- [Background] Bang YJ, Kim YW, Yang HK, Chung HC, Park YK, Lee KH, Lee KW, Kim YH, Noh SI, Cho JY, Mok YJ, Kim YH, Ji J, Yeh TS, Button P, Sirzen F, Noh SH; CLASSIC trial investigators. Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): a phase 3 open-label, randomised controlled trial. Lancet. 2012 Jan 28;379(9813):315-21. doi: 10.1016/S0140-6736(11)61873-4. Epub 2012 Jan 7. PMID 22226517
- [Background] Tsuburaya A, Yoshida K, Kobayashi M, Yoshino S, Takahashi M, Takiguchi N, Tanabe K, Takahashi N, Imamura H, Tatsumoto N, Hara A, Nishikawa K, Fukushima R, Nozaki I, Kojima H, Miyashita Y, Oba K, Buyse M, Morita S, Sakamoto J. Sequential paclitaxel followed by tegafur and uracil (UFT) or S-1 versus UFT or S-1 monotherapy as adjuvant chemotherapy for T4a/b gastric cancer (SAMIT): a phase 3 factorial randomised controlled trial. Lancet Oncol. 2014 Jul;15(8):886-93. doi: 10.1016/S1470-2045(14)70025-7. Epub 2014 Jun 18. PMID 24954805
- [Background] O'Connell MJ, Laurie JA, Kahn M, Fitzgibbons RJ Jr, Erlichman C, Shepherd L, Moertel CG, Kocha WI, Pazdur R, Wieand HS, Rubin J, Vukov AM, Donohue JH, Krook JE, Figueredo A. Prospectively randomized trial of postoperative adjuvant chemotherapy in patients with high-risk colon cancer. J Clin Oncol. 1998 Jan;16(1):295-300. doi: 10.1200/JCO.1998.16.1.295. PMID 9440756
- [Background] Chen S, Chen YB, Zhou ZW, Li W, Sun XW, Xu DZ, Li YF, Guan YX, Feng XY, Zhan YQ. No survival benefit from postoperative adjuvant chemotherapy after D2 radical resection for the patients with stage II gastric cancer. Am J Clin Oncol. 2011 Jun;34(3):309-13. doi: 10.1097/COC.0b013e3181dea94e. PMID 20838324
- [Background] Ji J, Liang H, Zhan Y, Liu Y, He Y, Ye Y, Sun Y, Huang C, Yan M, Shi Y, Wu A. [Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): Chinese subgroup analysis]. Zhonghua Wei Chang Wai Ke Za Zhi. 2014 Feb;17(2):133-8. Chinese. PMID 24577767
- [Background] Qu JL, Li X, Qu XJ, Zhu ZT, Zhou LZ, Teng YE, Zhang JD, Jin B, Zhao MF, Yu P, Liu YP. Optimal duration of fluorouracil-based adjuvant chemotherapy for patients with resectable gastric cancer. PLoS One. 2013 Dec 26;8(12):e83196. doi: 10.1371/journal.pone.0083196. eCollection 2013. PMID 24386161
- See also: cancer — https://www.nlm.nih.gov/medlineplus/cancer.html
- See also: stomach cancer — https://www.nlm.nih.gov/medlineplus/stomachcancer.html
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: S-1 — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0150863824&QV1=S1